CLINICAL TRIAL: NCT01846572
Title: Prevalence of Low Response to Clopidogrel in Patients After Acute Ischemic Stroke. The Bochumer CRISP Study
Brief Title: Clopidogrel Response in Acute Ischemic Stroke
Acronym: Bo-CRISP
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Saskia Meves, MD, Ruhr University of Bochum
Other Study IDs: RUB-Neuro-2013-clopi
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-04

CONDITIONS: Ischemic Stroke
Keywords: Stroke; Clopidogrel; Aggregometry; Antiplatelet therapy; Platelet function tests
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study was to determine the prevalence rate and risk factors for chemical laboratory clopidogrel low-response (CLR) in the acute phase after an ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* acute ischemic stroke
* admittance to stroke unit
* clopidogrel medication

Exclusion Criteria:

* no consent
* prior bleeding disorders
* severe liver disorders
* current gastrointestinal disorders
* congestive heart failure
* life-threatening malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an acute ischemic stroke admitted to our hospital and treated with clopidogrel
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2010-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Result of platelet function test | 1 day
  Aggregometry result of antiplatelet therapy

CONTACTS AND LOCATIONS:
Overall Officials: Saskia H Meves, MD, Principal Investigator — Ruhr University Bochum, Department of Neurology